CLINICAL TRIAL: NCT07150195
Title: Study on Proteomic and Microbiome Changes in Patients With Hepatic Encephalopathy (HE)
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Wenfang Chen
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Cirrhoses, Liver; Hepatic Encephalopathy (HE)
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal sample: Use a fecal collection tube to collect half of the tube. Collect the middle section of the fecal sample to avoid urine contamination. Mark the tube with the number, name, date and fecal score on the outside. Hand it over to the staff and immediately fresh divide it into 4 tubes, each tube about 500mg. Store it in a refrigerator at -80℃ and avoid freezing and thawing.
  2. Serum sample: Use a red-capped sterile blood collection tube (without additives) to draw 3ml of blood, and centrifuge to take 1.5ml of the supernatant. Evenly aliquot into 3 tubes for labeling, each tube approximately 500 μ l, and store in a -80 ° C refrigerator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver cirrhosis non-hepatic encephalopathy group (NHE group): Patients with liver cirrhosis aged ≥18 years, with normal blood ammonia; West-Haven classification 0, normal neurological signs, and normal neuropsychological tests; The patient agreed to participate and signed the informed consent form.
- Liver cirrhosis hepatic encephalopathy group (HE group）: Patients with liver cirrhosis aged 18 years or older, with elevated blood ammonia; Subclinical hepatic encephalopathy and West-Haven classification of grades 0, 1 to 4 HE, presenting with mental abnormalities such as personality and behavioral changes, and neurological abnormalities such as coma; Neurological signs are normal/flapping tremors can be elicited/positive neurological signs such as ankle clonus, and neuropsychological tests are abnormal; The patient/legal guardian agrees to participate and signs the informed consent form.

SUMMARY:
The objective of this observational study is to compare the differences in proteomics and gut microbiome between the liver cirrhosis group without hepatic encephalopathy and the hepatic encephalopathy group through proteomics and microbiome analysis, screen out the characteristic proteomics and microbiome of patients with hepatic encephalopathy, guide clinical diagnosis and treatment, and conduct in-depth research on the pathogenesis of hepatic encephalopathy. The main questions it aims to answer are:

Are there any differences in serum proteomes between patients with liver cirrhosis without hepatic encephalopathy and those with hepatic encephalopathy? If so, what are the main protein differences? There are differences in the fecal microbiome between patients with liver cirrhosis without hepatic encephalopathy and those with hepatic encephalopathy? If so, what are the main microbial differences?

This study will screen for the differences in proteomes and gut microbiomes between patients with liver cirrhosis without hepatic encephalopathy and those with hepatic encephalopathy, and identify the characteristic proteomes and microbiomes of patients with hepatic encephalopathy to guide clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

For the NHE (No Hepatic Encephalopathy) Group:

1. Aged between 18 and 85 years, inclusive.
2. Diagnosis of liver cirrhosis.
3. Normal blood ammonia level.
4. West-Haven Criteria grade 0 for Hepatic Encephalopathy.
5. Normal neurological signs.
6. Normal neuropsychological test results.
7. Willing to participate and provides written informed consent.

For the CHE (Covert Hepatic Encephalopathy) Group:

1. Aged between 18 and 85 years, inclusive.
2. Diagnosis of liver cirrhosis.
3. Elevated blood ammonia level.
4. Diagnosis of Covert Hepatic Encephalopathy (West-Haven Criteria grade 0 or I).

   * Grade 0: No personality or behavioral changes but abnormal neuropsychological tests.
   * Grade I: Mild cognitive impairment, lack of awareness, euphoria or anxiety, shortened attention span, or impaired performance of addition/subtraction.
5. Neurological signs are normal or mild asterixis (flapping tremor) may be elicited.
6. Neuropsychological tests are abnormal.
7. Willing to participate and provides written informed consent.

Exclusion Criteria:

1. Diagnosis of any malignant tumor.
2. History of treatment for any malignant tumor.
3. Presence of severe concomitant cardiac, pulmonary, cerebral, or renal diseases, or severe diabetic complications.
4. Use of antibiotics, prebiotics, probiotics, or proton pump inhibitors within the three months prior to enrollment.
5. Pregnancy, lactation, or puerperium.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population: A hospital-based cohort of adult patients (aged 18-85 years) with a confirmed diagnosis of liver cirrhosis, specifically recruited to form two distinct study groups based on the presence or absence of hepatic encephalopathy (HE) and blood ammonia levels.
  Sampling Method: Non-Probability Sample. Participants will be consecutively recruited from inpatient units. A purposive sampling strategy will be employed to ensure the successful enrollment of a sufficient number of participants in the Hepatic Encephalopathy (HE) group.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Microbiological and proteomic measurements | September 2025 - June 2026
  1. Microbiome Alpha Diversity (Shannon Index) Variable Name: Shannon Index Unit of Measure: Unitless (Shannon Index is a dimensionless quantity) Description: Alpha diversity assessed from 16S rRNA sequencing data using the Shannon Index, analyzed via QIIME.
  2. Relative Abundance of Specific Bacterial Taxa Variable Name: Relative Abundance Unit of Measure: % Description: The relative abundance of specific bacterial taxa, derived from 16S rRNA sequencing data analyzed using QIIME.
  3. Proteomic Abundance of Specific Proteins Variable Name: Protein Abundance Unit of Measure: Arbitrary Intensity Units Description: Abundance of specific proteins measured by mass spectrometry-based proteomic analysis.

SECONDARY OUTCOMES:
1.Demographic and Clinical Characteristics Assessment using Data Collection Forms 2.Cognitive Function Assessment using Mini-Mental State Examination (MMSE) 3.Laboratory Blood Parameters Measured by Standard Clinical Laboratory Assays | September 2025 - June 2026
  I. Participant Characteristics Sex (n) Height (m) Weight (kg) Body Mass Index, BMI (kg/m²) Disease Duration (months) Description: Data collected via questionnaire, medical record review, and physical measurement. BMI was calculated from height and weight.
  II. Cognitive Function Mini-Mental State Examination, MMSE Score (points, 0-30)
  III. Laboratory Parameters - Hematology Hemoglobin (g/dL) White Blood Cell Count (×10⁹/L) Platelet Count (×10⁹/L)
  IV. Laboratory Parameters - Coagulation Prothrombin Time (s)
  V. Laboratory Parameters - Liver Function and Metabolism Blood Ammonia (μmol/L) Serum Albumin (g/dL) Alanine Aminotransferase, ALT (U/L) Aspartate Aminotransferase, AST (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Wenfang Cheng, Study Director — Department of Gastroenterology, the First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Gastroenterology, the First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are currently undecided regarding sharing of Individual Participant Data (IPD). The primary reason for this uncertainty is to ensure full compliance with all regulatory obligations and to uphold the confidentiality commitments made to the study participants during the informed consent process.
  Therefore, sharing IPD would require further review and approval by the relevant Institutional Review Board (IRB)/Ethics Committee, and in some cases, may necessitate re-consenting participants, which is not always feasible.
  The investigators acknowledge the importance of data sharing for scientific progress. A final decision will be made following the completion of the study and publication of the primary results. The investigators will formally consult with the IRB/Ethics Committee and the data protection officers to determine if and how the data can be shared in a manner that is fully compliant with Chinese regulations and international standards for data privacy.

REFERENCES:
- [Result] Munk Lauridsen M, Jonasson E, Bajaj JS. Microbial Approaches to Treat and Prevent Hepatic Encephalopathy. Gastroenterol Clin North Am. 2025 Jun;54(2):429-451. doi: 10.1016/j.gtc.2024.12.006. Epub 2025 Jan 23. PMID 40348497
- [Result] Engelmann C. Rethinking hepatic encephalopathy: Gut microbes, neurotoxins and the therapeutic horizon. J Hepatol. 2025 Aug;83(2):601-603. doi: 10.1016/j.jhep.2025.04.036. Epub 2025 May 27. No abstract available. PMID 40436647
- [Result] Li S, Xu Z, Diao H, Zhou A, Tu D, Wang S, Feng Y, Feng X, Lai Y, Yang S, Tang B. Gut microbiome alterations and hepatic encephalopathy post-TIPS in liver cirrhosis patients. J Transl Med. 2025 Jul 4;23(1):745. doi: 10.1186/s12967-025-06774-y. PMID 40615853
- [Result] Mancini A, Campagna F, Amodio P, Tuohy KM. Gut : liver : brain axis: the microbial challenge in the hepatic encephalopathy. Food Funct. 2018 Mar 1;9(3):1373-1388. doi: 10.1039/c7fo01528c. Epub 2018 Feb 27. PMID 29485654
- [Result] Stengel S, Stallmach A, Richter K, Landrock A, Hampe J, Bruns T. Serum metabolic signatures in patients with overt hepatic encephalopathy. J Hepatol. 2017 Nov;67(5):1114-1115. doi: 10.1016/j.jhep.2017.06.030. Epub 2017 Jul 6. No abstract available. PMID 28690175

DOCUMENTS (1):
  • Informed Consent Form (2025-08-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT07150195/ICF_000.pdf